CLINICAL TRIAL: NCT00507091
Title: A Phase I Open Label Study to Asses the Safety and Tolerability of ZD6474 (Vandetanib)in Combination With Irinotecan, 5-Fluorouracil and Leucovorin (FOLFIRI) as First or Second Line Therapy in Patients With Metastatic Colorectal Adenocarcinoma.
Brief Title: Phase I Irinotecan, 5-Fluorouracil and Leucovorin Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00038
Record Dates: First submitted 2007-07-10; First posted 2007-07-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic; Colorectal; Adenocarcinoma
Keywords: ZD6474; Irinotecan; 5-Fluorouracil; Leucovorin; colorectal
MeSH Terms: conditions — Neoplasm Metastasis; Adenocarcinoma | interventions — vandetanib; Irinotecan; Fluorouracil; Leucovorin

ARMS (2):
- ZD6474 (vandetanib) 100mg (Experimental)
  Interventions: Drug: ZD6474 (vandetanib) 100mg; Drug: Irinotecan; Drug: 5-Fluorouracil; Drug: Leucovorin
- ZD6474 (vandetanib) 300mg (Experimental)
  Interventions: Drug: Irinotecan; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: ZD6474 (vandetanib) 300mg

INTERVENTIONS:
Drug: ZD6474 (vandetanib) 100mg — once daily oral tablet
  Other Names: ZACTIMA™
  Arms: ZD6474 (vandetanib) 100mg
Drug: Irinotecan — intravenous infusion
  Other Names: Camptosar®
Drug: 5-Fluorouracil — intravenous infusion
  Other Names: 5-FU
Drug: Leucovorin — intravenous infusion
Drug: ZD6474 (vandetanib) 300mg — once daily oral tablet
  Other Names: ZACTIMA™
  Arms: ZD6474 (vandetanib) 300mg

SUMMARY:
A Phase I open label study to asses the safety and tolerability of ZD6474 in combination with Irinotecan, 5-Fluorouracil and Leucovorin (FOLFIRI) as first or second line therapy in patients with metastatic colorectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed metastatic colorectal adenocarcinoma
2. Not amenable to surgery or radiation therapy
3. Eligible for first or second line chemotherapy

Exclusion Criteria:

1. Brain metastases or spinal compression
2. Last prior chemotherapy discontinued within 4 weeks before start
3. Last dose radiotherapy within 4 weeks of start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-08; Primary Completion 2006-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Establish the safety & efficacy of ZD6474 w/5-fluorouracil,leucovorin & oxaliplatin to patients with advanced colorectal adenocarcinoma, by assessment of AEs, vital signs, clinical chemistry, hematology, urinalysis, ECG and physical examinations | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Research Site, Ghent, Belgium
- United Kingdom (2):
  - Research Site, Belfast
  - Research Site, Manchester

REFERENCES:
- [Background] Saunders MP, Wilson R, Peeters M, Smith R, Godwood A, Oliver S, Van Cutsem E. Vandetanib with FOLFIRI in patients with advanced colorectal adenocarcinoma: results from an open-label, multicentre Phase I study. Cancer Chemother Pharmacol. 2009 Sep;64(4):665-72. doi: 10.1007/s00280-008-0914-4. Epub 2009 Jan 29. PMID 19184020
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1426&filename=CSR-D4200C00038.pdf
- See also: CSR-D4200C00038.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1426&filename=CSR-D4200C00038.pdf